CLINICAL TRIAL: NCT01479153
Title: Comparison of Subclavian, Femoral and Internal Jugular Venous Catheterization in Term of Complications in the Intensive Care Unit: a Randomized Controlled Trial
Brief Title: Venous Site for Central Catheterization
Acronym: 3SITES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ID RCB 2010-A00813-36
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2015-07

CONDITIONS: Critical Care; Catheterization; ICU
Keywords: Central venous catheterization; Major complications; Internal Jugular; Femoral; Subclavian
MeSH Terms: interventions — Catheterization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Subclavian catheterization (Active Comparator)
  Interventions: Procedure: Randomization of the site for catheterization
- Internal Jugular catheterization (Active Comparator)
  Interventions: Procedure: Randomization of the site for catheterization
- Femoral Catheterization (Active Comparator)
  Interventions: Procedure: Randomization of the site for catheterization

INTERVENTIONS:
Procedure: Randomization of the site for catheterization — Ultra-sound guided insertion strongly recommended

SUMMARY:
Central venous catheters are needed in the critical care setting to administer drugs. Three sites are available to gain vascular access: subclavian, internal jugular and femoral. Each site has complications, but there is no randomized controlled study which compared the 3 sites.

The investigators hypothesis is that subclavian catheterization reduces the risk of major complications compared to internal jugular or femoral.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted in the Intensive Care Unit
* Requiring Central Venous Catheterization

Exclusion Criteria:

* Patients with only one site available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3471 (Actual)
Dates: Start 2011-10; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Major complications including catheter-related bloodstream infection | From central catheter insertion to 48-h after removal
  Catheter-related bloodstream infection: (positive catheter-tip quantitative culture plus positive peripheral blood culture(s))

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Parienti, MD, PhD, Principal Investigator — CHU CAEN
Locations (5):
- France (5):
  - Medical Intensive Care Unit, CHU Caen, Caen
  - Surgical Intensive Care Unit, CHU Caen, Caen
  - Medical Intensive Care Unit, Cochin, AP-HP, Paris
  - Médical Intensive Care Unit, Lariboisière, AP-HP, Paris
  - Polyvalent Intensive Care Unit, Mémorial France Etats-Unis, Saint-Lô

REFERENCES:
- [Result] Parienti JJ, Mongardon N, Megarbane B, Mira JP, Kalfon P, Gros A, Marque S, Thuong M, Pottier V, Ramakers M, Savary B, Seguin A, Valette X, Terzi N, Sauneuf B, Cattoir V, Mermel LA, du Cheyron D; 3SITES Study Group. Intravascular Complications of Central Venous Catheterization by Insertion Site. N Engl J Med. 2015 Sep 24;373(13):1220-9. doi: 10.1056/NEJMoa1500964. PMID 26398070
- [Result] Pages J, Hazera P, Megarbane B, du Cheyron D, Thuong M, Dutheil JJ, Valette X, Fournel F, Mermel LA, Mira JP, Daubin C, Parienti JJ; 3SITES Study Group. Comparison of alcoholic chlorhexidine and povidone-iodine cutaneous antiseptics for the prevention of central venous catheter-related infection: a cohort and quasi-experimental multicenter study. Intensive Care Med. 2016 Sep;42(9):1418-26. doi: 10.1007/s00134-016-4406-4. Epub 2016 Jun 16. PMID 27311311
- [Derived] Iachkine J, Buetti N, de Grooth HJ, Briant AR, Mimoz O, Megarbane B, Mira JP, Valette X, Daubin C, du Cheyron D, Mermel LA, Timsit JF, Parienti JJ. Development and validation of a multivariable model predicting the required catheter dwell time among mechanically ventilated critically ill patients in three randomized trials. Ann Intensive Care. 2023 Jan 16;13(1):5. doi: 10.1186/s13613-023-01099-9. PMID 36645531
- [Derived] Iachkine J, Buetti N, de Grooth HJ, Briant AR, Mimoz O, Megarbane B, Mira JP, Ruckly S, Souweine B, du Cheyron D, Mermel LA, Timsit JF, Parienti JJ. Development and validation of a multivariable prediction model of central venous catheter-tip colonization in a cohort of five randomized trials. Crit Care. 2022 Jul 7;26(1):205. doi: 10.1186/s13054-022-04078-x. PMID 35799302